CLINICAL TRIAL: NCT02956174
Title: Posterior CAD/CAM Cobalt-chromium Alloy Single Crowns: 4-year Prospective Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Fernando Zarone, Full Professor, Federico II University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FZ_Co-Cr_2016
Record Dates: First submitted 2016-10-30; First posted 2016-11-07 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-11

CONDITIONS: Single Tooth Lost

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Co-Cr single crown (Experimental): Co-Cr single crown
  Interventions: Device: Co-Cr single crown; Other: Periodontal parameters
- Contralateral sound tooth (Active Comparator): Contralateral sound tooth
  Interventions: Other: Periodontal parameters

INTERVENTIONS:
Device: Co-Cr single crown
  Arms: Co-Cr single crown
Other: Periodontal parameters

SUMMARY:
Objectives - To evaluate the 4-year clinical outcomes of ceramic veneered Computer Aided Design/Computer Aided Manufacturing (CAD/CAM) Co-Cr single crowns supported by natural teeth in posterior regions.

Material and methods - Eighty-nine patients were provided with 120 ceramic veneered CAD/CAM Co-Cr single crowns replacing either premolars and molars. Specific inclusion criteria were needed and tooth preparations were standardized and performed by 2 expert prosthodontists. CAD/CAM Co-Cr frameworks were fabricated and veneered with ceramics. The restorations were cemented using a eugenol-free zinc oxide luting agent. The patients were recalled after 1, 6, 12, 24, 36 and 48 months. The survival and success of the restorations were evaluated. The technical and esthetic outcomes were examined using the United States Public Health Service criteria. The biologic outcomes were analyzed at abutment and contralateral teeth and descriptive statistics were performed.

ELIGIBILITY:
Inclusion criteria:

* good general health
* American Society of Anesthesiologists (ASA) ASA I or ASA II condition; periodontal health
* Angle class I occlusal relationship
* minimum of 10 couples of opponent teeth
* good oral hygiene
* no evident signs of parafunctions and/or temporomandibular disorders.
* periodontal health of abutment teeth (absence of tooth mobility, absence of furcation involvement);
* proper positioning of abutment teeth in the dental arch (tooth axis adequate for a SC)
* sufficient occlusal-cervical height of the clinical crown of abutment teeth (≥ 4 mm) for the retention of a SC
* vital or endodontically treated to a clinically sound state abutment teeth;
* abutment teeth opposing natural teeth.

Exclusion criteria:

* high caries activity
* presence of periodontal disease on the abutment tooth
* occlusal-cervical height of the abutment tooth < 4 mm
* reduced interocclusal distance or supraerupted opposing teeth
* unfavorable crown-to-root ratio
* severe were facets, clenching and/or bruxism
* presence of removable partial dentures (RPDs)
* pregnancy or lactation
* alcohol and/or drug addiction

Ages: 21 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2012-05; Primary Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Survival percentage | 4 years
  Kaplan Meier analysis of survival of the prostheses